CLINICAL TRIAL: NCT05142020
Title: Study on Early Screening Biomarkers of Gestational Diabetes Mellitus and Its Related Pathogenesis
Brief Title: Biomarkers for Early Screening of Gestational Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: Early Screening of GDM
Record Dates: First submitted 2021-06-13; First posted 2021-12-02 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Gestatiaonl Diabetes Mellitus; Early Pregnancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, plasma, serum, urine, tissue (placenta and umbilical cord)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GDM group: Specimen collection and clinical follow-up
- Control group: Specimen collection and clinical follow-up

SUMMARY:
Gestational Diabetes Mellitus (GDM) refers to the abnormal glucose metabolism first detected during pregnancy. It is estimated that approximately 7% of pregnant women worldwide and their offspring are affected by GDM. The incidence of GDM in China is as high as 18.9%. A number of studies have shown that GDM complicates 3%-25% of pregnancies and poses serious health and life threats to the mother and child. In fact, due to the lack of physical activity during pregnancy and the decrease of insulin sensitivity compared with non-pregnancy, the optimal time for intervention has long been lost until the diagnosis of GDM in the second trimester. However, it is a pity that no authoritative screening method for GDM in early pregnancy has been established, and the pathogenesis of GDM is still unclear. This study intend to search for biomarkers used for screening of GDM in early pregnancy and explore the pathogenesis of GDM, so as to provide new ideas for prevention measures and treatment targets of GDM.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age: 20-49 years
* Plan to have routine prenatal examinations and give birth in the research center
* Willing to cooperate with the hospital to follow up

Exclusion Criteria:

* Have diseases that affect metabolic function or even threaten the life of the mother and fetus before pregnancy, such as diabetes, hypertension, heart disease, liver and kidney diseases, thyroid diseases, autoimmune diseases, malignant tumors, AIDS, etc.
* Fetus has a known deformity or genetic defects
* Incomplete clinical data

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This project intends to recruit pregnant women who go to the research center for routine prenatal examination and OGTT screening.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Significantly different metabolites at 8-10 gestational weeks | Gestatioanl weeks: 8-10 weeks
  Metabolomics are used to screen out significant different metabolites. Specific metabolites indicators will be given based on the results of preliminary experiments. The changes of biomarkers are observed at different gestational weeks.
Significantly different metabolites at 16-18 gestational weeks | Gestatioanl weeks: 16-18 weeks
  Metabolomics are used to screen out significant different metabolites. Specific metabolites indicators will be given based on the results of preliminary experiments. The changes of biomarkers are observed at different gestational weeks.
Significantly different metabolites at 24-26 gestational weeks | Gestatioanl weeks: 24-26 weeks
  Metabolomics are used to screen out significant different metabolites. Specific metabolites indicators will be given based on the results of preliminary experiments. The changes of biomarkers are observed at different gestational weeks.
Significantly different metabolites at 32-34 gestational weeks | Gestatioanl weeks: 32-34 weeks
  Metabolomics are used to screen out significant different metabolites. Specific metabolites indicators will be given based on the results of preliminary experiments. The changes of biomarkers are observed at different gestational weeks.
Significantly different proteins at 8-10 gestational weeks | Gestatioanl weeks: 8-10 weeks
  Proteomics are used to screen out significant different proteins. Specific proteins indicators will be given based on the results of preliminary experiments. The changes of biomarkers are observed at different gestational weeks.
Significantly different proteins at 16-18 gestational weeks | Gestatioanl weeks: 16-18 weeks
  Proteomics are used to screen out significant different proteins. Specific proteins indicators will be given based on the results of preliminary experiments. The changes of biomarkers are observed at different gestational weeks.
Significantly different proteins at 24-26 gestational weeks | Gestatioanl weeks: 24-26 weeks
  Proteomics are used to screen out significant different proteins. Specific proteins indicators will be given based on the results of preliminary experiments. The changes of biomarkers are observed at different gestational weeks.
Significantly different proteins at 32-34 gestational weeks | Gestatioanl weeks: 32-34 weeks
  Proteomics are used to screen out significant different proteins. Specific proteins indicators will be given based on the results of preliminary experiments. The changes of biomarkers are observed at different gestational weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Danqing Chen, Hangzhou, Zhejiang, China